CLINICAL TRIAL: NCT00945113
Title: A Pilot Randomised Controlled Trial of the Effectiveness of Intensive Group Speech and Language Therapy as a Treatment for Older Children Who Stammer
Brief Title: Pilot: Group Therapy for Children Who Stammer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Collaborators: University of Newcastle Upon-Tyne (Other); North Tyneside Primary Care Trust (Unknown); Northumberland Care Trust (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: 4565
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Stammering
Keywords: pilot; stammer; stutter; children; randomised controlled trial; RCT; Speech and Language Therapy; Stuttering
MeSH Terms: conditions — Stuttering; Communication Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): attendance at one-week speech therapy group
  Interventions: Behavioral: One-week speech therapy group

INTERVENTIONS:
Behavioral: One-week speech therapy group — One-week cross-district speech therapy group for older children (aged 8 to 15) who stammer

SUMMARY:
The aim of the study is to answer the question: Is a large-scale research study of the effectiveness of group speech and language therapy (SALT) for young people who stammer possible?

The study will look at the issues involved in setting up a large-scale investigation of treatment for young people who stammer. It will inform the investigators whether larger studies would be possible and give some early-stage information on the effectiveness of group SALT for these young people. The findings will pave the way for building and testing out treatment programmes where there will be clear positive benefit for young people who stammer and their families.

To answer the research question, the study will tell the investigators (a) how easy/difficult it was to get people to take part, (b) young people and parents'/carers' views on taking part and (c) whether the assessments were able to pick up changes in speech and attitudes towards stammering reported by the young people and their carers.

Sufficient numbers of participants were not recruited to carry out the intended rehearsal pilot RCT study design.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8;0 years and 15;11 years at 20.07.09
* Currently in treatment, on review or on waiting list for treatment.
* Has had an initial NHS Speech and Language Therapy assessment by Newcastle, Northumberland or North Tyneside Speech and Language Therapy service.
* Has a diagnosis of stammering.
* Has sufficient understanding of spoken (English) language to score at or above the 16th percentile on the Understanding Linguistic Concepts subtest of the CELF-4UK assessment.
* Available to attend treatment for the whole week of 20th July 2009
* Available to attend treatment for the whole week of 24th August 2009

Exclusion Criteria:

* Diagnosis of Attention and/or Hyperactivity Disorders
* Diagnosis of moderate or severe general learning difficulties
* Diagnosis of moderate or severe receptive and/or pragmatic language difficulties
* Parent/carer for whom an interpreter would be required

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Overall Assessment of the Speaker's Evaluation of Stuttering (OASES) score | July 2009 week 2, July 2009 week 4, October 2009 week 4

CONTACTS AND LOCATIONS:
Overall Officials: Lucy E Paterson, MA, BSc, Principal Investigator — Newcastle upon Tyne NHS Hospitals Foundation Trust
Locations (1):
- Newcastle-upon-Tyne Hospitals NHS Trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom